CLINICAL TRIAL: NCT05379361
Title: Program Development Study for Developing Emotional Intelligence for Nursing Students
Brief Title: Program Development Study for Emotional Intelligence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, NİL KÜÇÜK YÜCEYURT, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IUC-FNHF
Record Dates: First submitted 2022-05-11; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Emotional Intelligence; Nursing; Education; Nurse's Role
Keywords: Emotional intelligence; Program Development; Students; Nursing; Education

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Emotional Intelligence Intervention Group (Experimental): Nursing students, whose Emotional Intelligence skills were aimed to be developed, formed the intervention group.
  Interventions: Behavioral: Emotional Intelligence Development Program
- Environmental Awareness Educational Group (Placebo Comparator): It is a group created to eliminate the risk of interaction about the intervention made due to the fact that nursing students are studying in the same semester and at the same faculty. Different from the intervention group, the students selected for this group were trained on environmental awareness, which is not related to Emotional Intelligence concepts and skills.
  Interventions: Behavioral: Plasebo Training Group
- No Intervention: Control Group (No Intervention): The control group consisted of the students who continued their nursing education and did not have any intervention or application for the development of emotional intelligence skills.

INTERVENTIONS:
Behavioral: Emotional Intelligence Development Program — It is a training program that was developed in line with the literature and preliminary research results and includes the bar-on emotional intelligence sub-dimensions.
  Arms: Emotional Intelligence Intervention Group
Behavioral: Plasebo Training Group — It is a training program that was developed in line with the literature and includes the environmental awareness skills education.
  Arms: Environmental Awareness Educational Group

SUMMARY:
For qualified nursing care, emotional intelligence skills of nurses should be developed during their vocational training. This research was carried out in order to develop and evaluate the Emotional Intelligence Training Program based on the Bar-On Emotional Intelligence Model for nursing students in line with Demirel's program development model.

DETAILED DESCRIPTION:
The experiment was planned in a randomized controlled experimental design with placebo, control group (pretest-posttest control pattern), blind technique. It is a research with a mixed pattern, since the individual in-depth interview method, one of the qualitative research methods, is also used in the research together with quantitative methods. The research was carried out with first-year nursing faculty students (N: 250) of a university.

The Emotional Intelligence training program created and was applied to the experimental group in the specified period. In order to minimize the risk of interaction, a different training program was simultaneously applied to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* The average score of the students on the emotional intelligence scale is in the range of 1-4 points.
* Willingness to participate in the study

Exclusion Criteria:

* Have received or receiving professional psychological or psychiatric support

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Emotional Intellligence Skills | Baseline (Before Education Program, posttest (2 weeks after education program ended)
  Bar-On Emotional Intelligence Scale

SECONDARY OUTCOMES:
Training Program Evaluation Questionnaire | Baseline
  Evaluation of the effectiveness of the training program carried out as an initiative.

CONTACTS AND LOCATIONS:
Overall Officials: Nil Küçük Yüceyurt, PhD, Study Chair — Istanbul Univesity Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuceyurt NK, Kaya H. Program development study focusing on emotional intelligence skills of nursing students: randomized controlled trial. BMC Nurs. 2025 Jul 7;24(1):859. doi: 10.1186/s12912-025-03491-1. PMID 40624641